CLINICAL TRIAL: NCT05106868
Title: Acupuncture for Patients With Major Depressive Disorder: Study Protocol of a Randomized Controlled Trial
Brief Title: Acupuncture for Patients With Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Di Qin, Professor, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-1273
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Major Depressive Disorder
Keywords: acupuncture; major depressive disorder; randomized controlled trial
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- acupuncture (Experimental): 5 sessions of acupuncture per week for 4 weeks. In each session, acupuncture will be applied bilaterally on acupoints. We will use transcutaneous electric acupoints stimulation (HANS; Han's acupoints nerve stimulator, HANS-200, Nanjing, China) to stimulate the acupoints. Each session will last 30 minutes.
  Interventions: Device: acupuncture
- sham acupuncture (Sham Comparator): 5 sessions of sham acupuncture per week for 4 weeks. In each session, acupuncture will be applied bilaterally on non-acupoints. We will use transcutaneous electric acupoints stimulation (HANS; Han's acupoints nerve stimulator, HANS-200, Nanjing, China) to stimulate the non-acupoints. Each session will last 30 minutes.
  Interventions: Device: acupuncture
- waiting-list (No Intervention)

INTERVENTIONS:
Device: acupuncture — Acupuncture is a form of alternative medicine and a component of traditional Chinese medicine (TCM) in which thin needles are inserted into the acupoints on body to treat diseases.
  Arms: acupuncture; sham acupuncture

SUMMARY:
Several studies investigating acupuncture for major depressive disorder (MDD) have been carried out. However, investigators found the results were in high heterogeneity and poor methodological quality. Thus, investigators intend to provide high quality of the effectiveness and safety of acupuncture for MDD.

ELIGIBILITY:
Inclusion Criteria:

1. Right-handed participants aged between 18 to 60 years;
2. participants diagnosed with mild to moderate major depressive disorder(MDD), and meet the diagnostic criteria of mild to moderate MDD according to the Diagnostic and Statistical Manual of Mental Disorders (Fifth Edition (DSM-5);
3. participants with score of HAMD-24 between 8 to 35;
4. participants without anti-depressive medication more than 3 months;
5. participants willing to comply with the study protocol;
6. participants willing to sign informed consent form.

Exclusion Criteria:

1. participants with severe medical visceral condition and chronic diseases, such as hypertension, coronary heart disease, hyperthyroidism, hypothyroidism or diabetes and other endocrine system diseases;
2. participants with brain organic diseases: such as birth injury, trauma, encephalitis, tumor, etc.;
3. participants with Peripheral nerve and muscular system diseases;
4. participants with severe anxiety, obsessive-compulsive disorder, or a history of mania or hypomania;
5. Recently taken drugs that may cause mood disorders;
6. Severe bleeding tendency, allergic constitution and skin disease patients;
7. pregnant or lactation women;
8. Persons with visual and hearing disabilities;
9. Participants with pacemakers, deep brain stimulators, vagus nerve stimulators, metal internal fixators, etc
10. participate in other clinical trials at the same time

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
score of Hamilton Depression Rating Scale-24 | change from baseline to 4 weeks after intervention, after follow-up(4 week)
  Reduction in the severity of depression, measured at the end of the intervention primarily as a continuous variable on the Hamilton Depression Rating Scale (HAMD)-24

SECONDARY OUTCOMES:
score of self-rating depression scale | baseline, after intervention(4 week), after follow-up(4 week)
  Reduction in the severity of depression, measured at the end of the intervention primarily as a continuous variable on self-rating depression scale (SDS)
score of Hamilton Anxiety Rating Scale | baseline, after intervention(4 week) , after follow-up(4 week)
  Reduction in the severity of depression, measured at the end of the intervention primarily as a continuous variable on Hamilton Anxiety Rating Scale (HAMA)
score of Social Disability Screening Schedule | baseline, after intervention(4 week) , after follow-up(4 week)
  change of score of Social Disability Screening Schedule (SDSS)
score of Pittsburgh sleep quality index (PSQI) | baseline, after intervention(4 week) , after follow-up(4 week)
  change of score of Pittsburgh sleep quality index (PSQI)
motor threshold (MT) | baseline, after intervention(4 week) , after follow-up(4 week)
  motor threshold (MT) measured by Brain Ultimate Combined with MEB-2312 EMG/evoked potentiometer
Intra-cortical facilitation (ICF) | baseline, after intervention(4 week) , after follow-up(4 week)
  Intra-cortical facilitation (ICF) measured by Brain Ultimate Combined with MEB-2312 EMG/evoked potentiometer
cortical resting period (CSP) | baseline, after intervention(4 week) , after follow-up(4 week)
  cortical resting period (CSP) measured by Brain Ultimate Combined with MEB-2312 EMG/evoked potentiometer [Time Frame: baseline, after intervention(4 week), after follow-up(4 week)]
intra-cortical inhibition (ICI) | baseline, after intervention(4 week) , after follow-up(4 week)
  intra-cortical inhibition (ICI) measured by Brain Ultimate Combined with MEB-2312 EMG/evoked potentiometer
IAPS Evoked Event-related Potentials (ERP) | baseline, after intervention(4 week), after follow-up(4 week)
  IAPS Evoked Event-related Potentials (ERP)
Evoked Event-related Potentials (ERP) in TMS-EEG | baseline, after intervention(4 week), after follow-up(4 week)
  Evoked Event-related Potentials (ERP) in TMS-EEG
Adverse events | during intervention(4 week)
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, Study Chair — Institute of Science and Technology Development, Sichuan University

IPD SHARING:
Plan to Share IPD: No